CLINICAL TRIAL: NCT04815837
Title: An Evidence-based Knowledge Transfer Program Promoting Human Papillomavirus (HPV) Vaccination Among Men Who Have Sex With Men in Hong Kong
Brief Title: An Online Intervention Promoting HPV Vaccination Among Chinese MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KPF18HLF22
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Vaccine Refusal
Keywords: HPV vaccination
MeSH Terms: conditions — Vaccination Refusal | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants received the following interventions:
  1. Viewing a video promoting Human Papillomavirus (HPV) vaccination
  2. Receiving discount coupons
  3. Visiting the project webpage
  4. Receiving follow-up reminders
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — 1. Viewing a video promoting Human Papillomavirus (HPV) vaccination: participants will watch a 5-minute online video promoting MSM's uptake of HPV vaccination. In the video, a peer MSM discussed about the risk of contracting HPV and having anal cancers among MSM, severe consequences of HPV-related diseases, as well as the benefits of HPV vaccination. He also demonstrated the procedures of taking up HPV vaccination in the collaborative private clinics, which portrayed caring, privacy guaranteed, and non-judgmental environment.
  2. Receiving the discount coupons: each participant will be given a discount coupon. By using the coupon, one can enjoy a 10% discount for taking up three doses of HPV vaccines at a collaborating private clinic.
  3. Visiting the project webpage: Participants can assess the project webpage by scanning the QR code on the discount coupon.
  4. Follow-up reminders: participants received five reminders at Month 1, 2, 4, 6, & 8.

SUMMARY:
Hong Kong Chinese speaking men who have sex with men completed a baseline survey, and then received an online intervention promoting uptake of Human Papillomavirus (HPV) vaccination. All participants are followed up by telephone 12 months after the completion of baseline survey.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate prevalence of uptake of Human Papillomavirus (HPV) vaccination after exposure to health promotion among men who have sex with men in Hong Kong within a 12-month project period.

Inclusion criteria are Hong Kong Chinese speaking males aged 18-45 years old and self-reported having had oral or anal intercourse with at least one man in the last six months. Those who have ever received HPV vaccination are excluded.

Participants are recruited through outreaching in gay venues, online advertisement and referral made by peers and non-governmental organization. With verbal informed consent, participants completed a baseline survey through telephone. They are then exposed to online interventions including: 1) watching an online video, 2) receiving a discount coupon to receive HPV vaccination at collaborative private clinics, 3) visiting the project webpage, and 4) receiving follow-up reminders 1, 2, 4, 6, and 8 months after the baseline survey.

All participants are followed up by telephone 12 months after the baseline survey to access the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese speaking males aged 18-45 years old and self-reported having had oral or anal intercourse with at least one man in the last six months

Exclusion Criteria:

* Have received any HPV vaccination

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on gender identity
Enrollment: 350 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Taking up at least one dose of Human Papillomavirus (HPV) vaccination in the past year | 12 months
  Participants report how many doses of HPV vaccines they have taken up in the past year.

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No